CLINICAL TRIAL: NCT04765085
Title: Study on the Clinical Efficacy and Change of Life Quality Through Using the Comprehensive Behavioral Intervention Treatment for Tics (CBIT)
Brief Title: Clinical Efficacy and Change of Life Quality Through Using the Comprehensive Behavioral Intervention Treatment for Tics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lacking of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sunjinhua
Record Dates: First submitted 2020-08-21; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Tic Disorders
Keywords: comprehensive behavioral intervention therapy; drug therapy; Psychosocial education
MeSH Terms: conditions — Tic Disorders | interventions — Aripiprazole; Tablets

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBIT Group (Experimental): Patients in this group would only receive the CBIT treatment.
  Interventions: Behavioral: comprehensive behavioral intervention therapy (CBIT)
- Drug therapy Group (Experimental): Patients in this group would only receive the drug therapy.
  Interventions: Drug: Aripiprazole 5Mg Oral Tablet

INTERVENTIONS:
Behavioral: comprehensive behavioral intervention therapy (CBIT) — Comprehensive behavioral intervention for tics is an extension of habit reversal training. It includes an expanded set of strategies, such as psycho-education about tic disorders, tic awareness training, competing response training, relaxation training, and functional analysis.
  According to the CBIT treatment manual (translated by sun Jinhua and Xu Wen, the author were Douglas W. woods et al., Oxford University Press, New York). The treatments consisted of 8 sessions for 10 weeks The first two phases were 1.5 hours, the last six stages were 1 hour.The treatment process was regularly supervised by a treatment supervisor.
  Arms: CBIT Group
Drug: Aripiprazole 5Mg Oral Tablet — Considering the patients with chronic tic disorder (chronic motor or vocal tic disorder or Tourette's disorder), aripiprazole was selected as a single drug with constant dose during the treatment. In case of extrapyramidal side effects, benhexol was given to reduce the extrapyramidal side effects, and the dosage and duration of medication were recorded
  Arms: Drug therapy Group

SUMMARY:
Study on the clinical efficacy and change of life quality through using the Comprehensive Behavioral Intervention Treatment for Tics (CBIT)

DETAILED DESCRIPTION:
This study tried to explore the clinical effect of comprehensive behavioral intervention therapy (CBIT) on tic symptoms and the effect of improving the quality of life in children with tic disorders;explore the optimal treatment plan for tic disorder by comparing the clinical efficacy of CBIT therapy, drug therapy, and psychosocial education; explore the feasibility of using quality of life as an evaluation index for functional recovery after tic disorder treatment;

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for chronic tic disorder or Tourette syndrome (TS) according to the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V), and has been diagnosed by two pediatric psychiatrists who are associate chief physicians or more;
* The age ranged from 9 to 16 years old;
* The total score of tic symptoms in the Yale global Tic Severity Scale (YGTSS) is 13-30;
* Childrens Webster's Intelligence Scale ≥ 85
* Co-morbid ADHD, but the drug treatment dose for ADHD is stable (the drug has been stabilized for more than 6 weeks), or no drug has been taken at the beginning and during the stud

Exclusion Criteria:

* There are brain organic diseases, metabolic diseases, psychiatric disorders, drug-induced involuntary movement and other extrapyramidal lesions;
* Habit reversal training and other behavioral treatments for more than 4 weeks;
* unwilling participants or disobedient subgroups in the study

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of Tic symptom severity before and after intervention | Baseline, the tenth week of treatment
  Tic symptom severity is estimated by Yale Global Tic Severity Scale Total Tic score. The YGTSS is a clinician-rated scale used to assess tic severity over the prior week. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics-scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from0 to 50. The Total Tic Score (YGTSS-TTS) was used in these analyses.Lower scores indicate improvement and higher scores indicate worsening.
  Reduction rate = (YGTSS total score before intervention - YGTSS total score after intervention) / YGTSS total score before treatment × 100%

SECONDARY OUTCOMES:
overall treatment response | The fifth week and the tenth week of treatment and three month after treatment end
  The overall treatment response is measured by CG-I. This is a repeated measurement variable.The CGI-I was used to measure overall treatment response. The scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse). We defined positive response as a score of 1 or 2 (much improved or very much improved).
life quality | The fifth week and the tenth week of treatment and three month after treatment end
  Pediatric Quality of Life Inventory (PedsQL) and Child Tourette's Syndrome Impairment Scale(CTIM) were used to assessed health-related QoL.This is a repeated measurement variable.
  PedsQL was a widely used 15-item measure assessed health-related QoL. Parents were asked to rate how often a particular item had been a problem during the past month using a 5-point Likert scale ranging from ''never a problem'' to ''almost always a problem." Total scores were linearly transformed to a scale of 0 to 100. Higher scores indicated better QoL. Four subscales measured physical, emotional, social, and school functioning.
  The CTIM-P is a 37-item parent-rated instrument that includes school, home, and social activities that may be impaired by their child's tics or a co-morbid problem (e.g., obsessive-compulsive symptoms, depressed mood, anxiety, oppositional/disruptive behavior, hyperactivity, inattentiveness).